CLINICAL TRIAL: NCT00960219
Title: D-amino Acid Oxidase Inhibition for NMDA Modulation in Schizophrenia
Brief Title: D-amino Acid Oxidase Inhibition (DAAOI-1) add-on Treatment for Chronic Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Hsien-Yuan Lane, M.D., Ph.D, Department of Psychiatry, China Medical University Hospital, Taichung, Taiwan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NSC-97-2314-B-039-006-MY3; NSC-97-2314-B-039-006-MY3
Record Dates: First submitted 2009-08-14; First posted 2009-08-17 (Estimated); Last update posted 2011-07-11 (Estimated); Status verified 2011-07

CONDITIONS: Schizophrenias; Psychoses; Psychotic Disorders; Schizophrenic Disorders
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Starch

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DAAOI-1 (Experimental)
  Interventions: Drug: D-amino acid oxidase inhibition (DAAOI-1)
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: D-amino acid oxidase inhibition (DAAOI-1) — 1g/day(500mg BID), oral, for 6 weeks
  Other Names: DAAOI-1
  Arms: DAAOI-1
Drug: placebo — 1# BID, oral, for 6 weeks
  Other Names: starch
  Arms: placebo

SUMMARY:
Adjuvant N-methyl-D-aspartic acid (NMDA)-enhancing agents, such as GlyT-1 inhibitors and NMDA-glycine site agonists have been demonstrated to be beneficial for chronic schizophrenia patients. The purpose of this study is to evaluate efficacy and safety of add-on treatment of an inhibitor of D-amino acid oxidase (DAAOI), DAAOI-1, in chronically stable schizophrenia patients who have been stabilized with antipsychotics.

DETAILED DESCRIPTION:
The etiology of schizophrenia remains unclear. Schizophrenia patients reveal positive symptoms, negative symptoms, and cognitive impairments. In addition to dopamine system hyperactivity, hypofunction of N-methyl-D-aspartate (NMDA) receptor plays a role in the pathophysiology of schizophrenia. Consequently, enhancing NMDA receptor neurotransmission has been regarded as a novel treatment approach. To date, several reported trials on adjuvant NMDA-enhancing agents, including glycine, D-amino acids (D-serine, D-alanine), and sarcosine (a glycine transporter I inhibitor), revealed beneficial but limited efficacy for positive and negative symptoms.

DAAOI-1 is a D-amino acid oxidase (DAAO) inhibitor which can elevate synaptic concentration of D-amino acids. The aim of this project is to examine the efficacy and safety of add-on treatment of DAAOI-1 in chronically stable schizophrenia patients who have been stabilized with antipsychotics.

In the study, 60 schizophrenic patients are recruited into the 6-week trial and randomly assigned into the two groups (1 gm/dDAAOI-1, or placebo) with a double-blind manner. Positive and Negative Syndrome Scale (PANSS), Scales for the Assessment of Negative symptoms (SANS), Global Assessment of Function (GAF), quality of life (QOL), Hamilton Depression rating scale 17(HAM-D 17), Clinical Global Impression(CGI)and side effects are evaluated every two weeks during the trial. Cognitive function ("7 domains of Measurement and Treatment Research to Improve Cognition in Schizophrenia" [MATRICS])are assessed at weeks 0 and 6. The efficacies of two groups are compared.

ELIGIBILITY:
Inclusion Criteria:

* Are physically healthy and have all laboratory assessments (including urine/blood routine, biochemical tests, and electrocardiograph) within normal limits
* Aged 18-65 year
* Fulfill the criteria of schizophrenia according to the Diagnostic and Statistical Manual, fourth edition (DSM-IV)
* Remain symptomatic but without clinically significant fluctuation and the antipsychotic doses are unchanged for at least 3 months
* Have a minimum baseline total score of 60 on the Positive and Negative Syndrome Scale (PANSS)
* Agree to participate in the study and provide informed consent

Exclusion Criteria:

* DSM-IV diagnosis of substance (including alcohol) abuse or dependence,
* DSM_IV diagnosis of mental retardation
* History of epilepsy, head trauma or CNS diseases
* History of epilepsy, head trauma or CNS diseases
* Pregnancy or lactation
* Inability to follow protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2009-04; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Total scores of PANSS, SANS, GAF, and QOL | week 0, 2, 4, 6.
Cognitive function | Week 0, 6
  MATRICS (Measurement and Treatment Research to Improve Cognition in Schizophrenia), including:1) speed of processing;(2) sustained attention; 3) working memory, verbal and nonverbal; 4) verbal learning and memory; 5) visual learning and memory; 6) reasoning and problem solving, and 7) social cognition

SECONDARY OUTCOMES:
The subscales of PANSS | week 0,2,4,6
Hamilton Depression rating scale 17(HAM-D 17) | Week 0, 2, 4, 6
Clinical Global Impression(CGI) | Week 0, 2, 4, 6

CONTACTS AND LOCATIONS:
Overall Officials: Hsien-Yuan Lane, M.D., Ph.D, Principal Investigator — Department of Psychiatry, China Medical University Hospital, Taichung, Taiwan
Locations (1):
- Department of Psychiatry, China Medical University Hospital, Taichung, Taiwan

REFERENCES:
- [Derived] Lane HY, Lin CH, Green MF, Hellemann G, Huang CC, Chen PW, Tun R, Chang YC, Tsai GE. Add-on treatment of benzoate for schizophrenia: a randomized, double-blind, placebo-controlled trial of D-amino acid oxidase inhibitor. JAMA Psychiatry. 2013 Dec;70(12):1267-75. doi: 10.1001/jamapsychiatry.2013.2159. PMID 24089054